CLINICAL TRIAL: NCT06952205
Title: Efficiency of Function-oriented Taping Application in Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Muhammed Fatih Kavak, Asst. Prof., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MFKavak-01
Record Dates: First submitted 2025-02-17; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain; Kinesiophobia
Keywords: Rigid taping; Functional taping
MeSH Terms: conditions — Low Back Pain; Kinesiophobia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- functional taping (Experimental): McKenzie exercises, Transcutaneous Electrical Nerve Stimulation (TENS), Hot Pack (HP) and pulsed ultrasound treatments were applied.To experimental group, functional taping were applied in addition of these treatments.
  Interventions: Other: Experimental group; Other: only exercises
- control group with only exercises (Active Comparator): McKenzie exercises, Transcutaneous Electrical Nerve Stimulation (TENS), Hot Pack (HP) and pulsed ultrasound treatments
  Interventions: Other: only exercises

INTERVENTIONS:
Other: Experimental group — McKenzie exercises, Transcutaneous Electrical Nerve Stimulation (TENS), Hot Pack (HP) and pulsed ultrasound treatments were applied.To experimental group, functional taping were applied in addition of these treatments.
  Arms: functional taping
Other: only exercises — McKenzie exercises, Transcutaneous Electrical Nerve Stimulation (TENS), Hot Pack (HP) and pulsed ultrasound treatments

SUMMARY:
Purpose of this study is to determine the efficiency of functional tape application to patients with acute or subacute low back pain. 40 patients with acute-subacute low back pain were divided into two groups: control and experimental group. To control group, McKenzie exercises, Transcutaneous Electrical Nerve Stimulation (TENS), Hot Pack (HP) and pulsed ultrasound treatments were applied. To experimental group, functional taping were applied in addition of these treatments. Range of Motion (ROM), Visual Analogue Scale (VAS), Tampa Scale of Kinesiophobia (TSK) and The Oswestry Disability Index (ODI) were evaluated preand post-treatment and datas were analyzed with statistical methods. In analysis; p value was accepted p<0,05 for t test and Mann Whitney U test process. In the measurements that compared the improvement of both groups, based on pre- and post-treatment evaluations; improvement in the experimental group was significantly higher in all of these parameters of ROM, VAS, TSK and ODI than in the control group (p<0,05). The use of functional rigid taping in patients with acute and subacute low back pain provided a statistically significant improvement in all measured values of patients and provide better results than the control group. However, there is a need for comparative new studies in order to measure the effectiveness of rigid taping in a more accurate way.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 20 and 65
* Being literate in Turkish
* Having lower back pain for less than 3 months
* Informed Consent Form for taping application to have been signed

Exclusion Criteria:

* Allergic reaction on the skin
* Hypertension, Type 2 diabetes mellitus (DM) and Presence of accompanying systemic disease other than hypercholesterolemia
* Not being able to communicate
* Using corsets and similar supports
* Having a body mass index > 30
* Use of antidepressant and myorelexan medication

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-23 (Actual)

PRIMARY OUTCOMES:
Range of Motion | through study completion, an average of 2 weeks.
  The flexion, extension, rotation, and lateral flexion range of motion of the lumbar region will be measured using a goniometer
Pain intensity | through study completion, an average of 2 weeks.
  The Visual Analog Scale (VAS) will evaluate low back pain by asking participants to mark their pain level on a 10 cm scale, where 0 indicates no pain and 10 indicates severe pain, based on their experience over the past week.
Degree of kinesiophobia | through study completion, an average of 2 weeks
  The Tampa Kinesiophobia Scale measures an individual's level of fear related to movement. Participants complete a 17-item questionnaire, indicating their fear and anxiety levels towards specific physical activities or movements. The scale uses a scoring system from 1 to 4 for each item, with a total score of up to 68. Higher scores indicate a higher level of kinesiophobia, while lower scores indicate less fear.
Disability Index | through study completion, an average of 2 weeks
  The Oswestry Disability Index (ODI) measures functional limitations in daily activities due to low back pain. The questionnaire consists of 10 sections, each assessing difficulties experienced by the participant due to pain. Participants rate each section from 0 to 5. The total score indicates the level of disability, with higher scores reflecting greater limitations in the individual's quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Uskudar Üniversity Physiotherapy and Rehabilitation Department, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No